CLINICAL TRIAL: NCT04515199
Title: Effectiveness of Telemedicine Use in Home Management of Adult Egyptian Mild COVID-19 Cases
Brief Title: Home Management of Adult Egyptian Mild COVID-19 Cases
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Tharwat Hegazy, Lecturer of Internal Medicine, Rheumatology and Clinical Immunology, Cairo University
Other Study IDs: Telemedicine in Mild COVID-19
Record Dates: First submitted 2020-08-07; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Telemedicine; Quality of Life; Safety Issues; Symptoms
Keywords: COVID19; Telemedicine; Home Isolation; Mild cases
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Keeping in mind the rising number of cases in Egypt and the strain they put on hospital infrastructure, the idea of home isolation and follow up for COVID 19 positive cases has been adopted in many countries and was approved by World Health Organization (WHO) and Egyptian Ministry of health (MOH).

Telehealth can help to mitigate this risk by minimizing the amount of face-to-face interactions. The WHO mentioned telemedicine among essential services in "strengthening the Health Systems Response to COVID-19" policy. The aim in this study is to study the effectiveness of telemedicine in managing mild COVID cases regarding isolation measures, symptoms, medications adherence, and reporting of red flags and side effects.

DETAILED DESCRIPTION:
Objectives:

* To assess the effectiveness of follow up of mild COVID-19 cases in home isolation
* To assess the applicability of telemedicine tools in the follow up of those patients and early identification of warning symptoms needing more intensive management measures.
* To assess the clinical characteristics for mild COVID-19 cases and post covid sequelae and the course of symptoms
* To assess the persistence of symptoms during follow up.
* To assess the quality of life during home management period.
* To assess cost-effectivenes of home isolation vs hospital admission in mild COVID-19 cases.

Study population & Sample size :

The study includes 400 Adult (18-65 years) Egyptian patients with mild COVID 19 diagnosed by PCR consented (oral consent) to home isolation to follow them.

Study Design:

Prospective observational study.

Methods:

• All patients will be subjected to thorough history and clinical examination. 400 adult mild COVID cases consented to home isolation to follow them by: phone calls, what's app, hot line for emergency, Triage sheet, zoom meetings.

Patients will be given brochures about home isolation (by Egyptian MOH), list of medications, plan of follow up.

1. Daily follow up for: fever chart, report any new symptoms or progression of previously present symptom or presence of red flags.
2. Blood samples will be obtained and CT chest will be done according to the usual protocol.
3. Patients will be followed for 3 months to detect post covid sequelae and the course of symptoms (and the persistence of any symptoms).
4. Questionnaire will be done to assess the patients' commitment to the advices and regulations of home isolation as well as forms to assess fatigue and the quality of life (36-Item Short Form Survey; SF-36).

ELIGIBILITY:
Inclusion Criteria:

1. No co-morbidities that necessitates hospital admission due to high risk for progression of the disease: Pregnancy, uncontrolled Diabetes, Chronic lung disease, Chronic kidney disease, Chronic liver disease, Serious heart diseases (arrythmia, Ischemic heart disease, uncontrolled hypertension), immunocompromised: prolonged use of corticosteroids and other immunosuppressive drugs/ organ transplantation/ HIV/ Immunodeficiency.
2. No fever (oral, below or equal 37.50 C )
3. No shortness of breath (Respiratory rate 12-20/min)
4. Oxygen saturation >= 96 %
5. CT chest: Normal
6. Labs: D-dimer<1000ng/ml, CPK< twice upper limit of normal, CRP<100, LDH<245, Ferritin<500, absolute lymphocytic count >0.8

Exclusion Criteria:

1. Moderate and severe cases not fulfilling the definition of mild cases.
2. Children and young < 18 years.
3. Age >65 years.
4. Presence of any of the previously mentioned comorbidities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 adult mild COVID cases consented to home isolation to follow them by: phone calls, what's app, hot line for emergency, Triage sheet, zoom meetings.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Percent of adherence to isolation measures | 3-6 months
  A checklist to check the percent of the patients who followed the advices for home isolation and will be validated
The incidence of symptoms and their duration | 3-6 months
  days

SECONDARY OUTCOMES:
Change in Short Form 35 (SF-36) Questionnaire | 3-6 months
  A validated questionnaire assessing function and quality of life for patients with pulmonary function issues
Cost- effectiveness of Home Isolation vs hospital admission in mild COVID-19 cases | 3-6 months
  We will measure the costs of home isolation vs hospital admission through collectin the expected costs if those mild cases have been admitted in the hospital as in the start of the crisis.
Identifying the duration of post-COVID-19 symptoms | 3-6 months
  Days
long-term respiratory complications | 3-6 months
  Interstitial lung disease diagnosed with a thoracic CT-scan

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim El Ebrashy, Professor, Principal Investigator — Internal Medicine Department, Faculty of Medicine, Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wynants L, Van Calster B, Collins GS, Riley RD, Heinze G, Schuit E, Bonten MMJ, Dahly DL, Damen JAA, Debray TPA, de Jong VMT, De Vos M, Dhiman P, Haller MC, Harhay MO, Henckaerts L, Heus P, Kammer M, Kreuzberger N, Lohmann A, Luijken K, Ma J, Martin GP, McLernon DJ, Andaur Navarro CL, Reitsma JB, Sergeant JC, Shi C, Skoetz N, Smits LJM, Snell KIE, Sperrin M, Spijker R, Steyerberg EW, Takada T, Tzoulaki I, van Kuijk SMJ, van Bussel B, van der Horst ICC, van Royen FS, Verbakel JY, Wallisch C, Wilkinson J, Wolff R, Hooft L, Moons KGM, van Smeden M. Prediction models for diagnosis and prognosis of covid-19: systematic review and critical appraisal. BMJ. 2020 Apr 7;369:m1328. doi: 10.1136/bmj.m1328. PMID 32265220
- [Background] Shi Y, Yu X, Zhao H, Wang H, Zhao R, Sheng J. Host susceptibility to severe COVID-19 and establishment of a host risk score: findings of 487 cases outside Wuhan. Crit Care. 2020 Mar 18;24(1):108. doi: 10.1186/s13054-020-2833-7. No abstract available. PMID 32188484
- [Background] Lee C, Chen D, Katz RL. Characteristics of nondepolarizing neuromuscular block: (I) post-junctional block by alpha-bungarotoxin. Can Anaesth Soc J. 1977 Mar;24(2):212-9. doi: 10.1007/BF03006234. PMID 139198